CLINICAL TRIAL: NCT06994715
Title: Effects of Acupressure Applied to Intensive Care Patients on Physiological Parameters, Pain, Sleep Quality, Anxiety and Perception of Nursing Presence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Özlem Canbolat, Gazi University, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-77082166-302.08.01-1229645
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Acupressure; Intensive Care Unit; Anxiety; Nursing Presence; Sleep Quality; Physiological Parameters
Keywords: Acupressure; intensive care unit; anxiety; nursing presence; sleep quality; physiological parameters
MeSH Terms: conditions — Anxiety Disorders; Sleep Initiation and Maintenance Disorders | interventions — Acupressure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Application group (Experimental): After the purpose of the study and the method of application are explained to the intensive care patients, the "Introductory Information Form", "Glasgow Coma Scale", "Visual Assessment Scale", "Physiological Parameters Assessment Form", "Richards-Campbell Sleep Scale", "Nursing Presence Scale" and "Spielberg State-Trait Anxiety Scale" will be applied. A total of 8 sessions of acupressure will be applied morning and evening for 2 days. The measurements will be repeated afterwards.
  Interventions: Other: Acupressure
- Placebo Group (Placebo Comparator): After the purpose of the study and the method of application are explained to the intensive care patients, the "Introductory Information Form", "Glasgow Coma Scale", "Visual Assessment Scale", "Physiological Parameters Assessment Form", "Richards-Campbell Sleep Scale", "Nursing Presence Scale" and "Spielberg State-Trait Anxiety Scale" will be applied. A total of 8 sessions of pseudo acupressure will be applied morning and evening for 2 days. Only light pressure will be applied without massage 2 cm to the side of the real points. The procedure will be performed with gloves. The measurements will be repeated afterwards.
  Interventions: Other: pseudo acupressure
- Control Group (No Intervention): No application will be made to the control group.

INTERVENTIONS:
Other: Acupressure — The patient will be placed in a suitable position (supine) or alternatively in a side-lying position, and the patient's privacy will be taken into account to determine the pressure points. The patient's own finger measurement will be taken into account when determining the pressure points. Acupressure points will be marked using a surgical marking pen. The pressure will be applied manually. The thumb will be used for this. Before applying direct pressure to the point, a light rubbing movement will be made for approximately 15 seconds on the point area to reduce tension and tissue sensitivity, to warm, relax and prepare. Approximately 2 minutes of pressure will be applied to each point in a circular manner. Each application will last approximately 18 minutes. The patient will be measured 9 times in total during 4 sessions.
  Arms: Application group
Other: pseudo acupressure — A pseudo acupressure will be applied to the patients in the supine or side-lying position. The researcher will perform this application by wearing gloves. Wearing gloves will reduce the therapeutic interaction with the patient. Since applying pressure or circular rubbing movements to patients may enter the area where other meridians pass and create a different effect, it will be waited for 2 minutes without applying any pressure or rubbing movements on the bone protrusions where the meridian does not pass and where there are no active pressure points. The application will be determined to be approximately 2 cm away from the acupressure points. The application will again be done manually with the thumb. Each application will take approximately 18 minutes. 4 sessions of application and a total of 9 measurements will be made to the patients.
  Arms: Placebo Group

SUMMARY:
This study will be conducted in a randomized controlled experimental design to examine the effects of acupressure applied to patients treated in the intensive care unit on physiological parameters, pain, sleep quality, anxiety and perception of nurse presence. The study will be conducted with 60 patients (20 intervention, 20 placebo, 20 control groups) treated in the 2nd stage Intensive Care Unit of an University Hospital between May 2025 and January 2026. Acupressure will be applied to the intervention group for 2 days, morning and evening, for four sessions. For four sessions, pseudo acupressure will be used on the placebo group for 2 days, morning and evening. No application will be made to the control group. The data collection tools in the study are the Patient Identifier Information Form, Glasgow Coma Scale (GCS), Visual Assessment Scale (VAS), Physiological Parameter Assessment Form, Richards-Campbell Sleep Scale, Spielberg State-Trait Anxiety Inventory, and Nurse Presence Scale (PONS).

ELIGIBILITY:
Inclusion Criteria:

* Have received intensive care treatment for at least 48 hours,
* Are 18 years of age or older,
* Have a Glasgow Coma Scale score of >13,
* Can speak and write in Turkish,
* Have no psychiatric diagnosis,
* Have no communication problems,
* Have a VAS score of ≥1,
* Have a mean arterial pressure of ≥65,
* Have SpO2 of ≥85.

Exclusion Criteria:

Have previously received acupressure treatment,

* Have ulcers, necrotic tissue and signs and symptoms of infection at the points where pressure will be applied,
* Have used antihypertensives, beta-blockers and similar medications,
* Have sedation,
* Have respiratory support from the device,
* Have inotropic treatment (dopamine, steradin and others),
* Have analgesic treatment in their routine treatment will not be included in the study.

Patients who were discharged during the study,

* Patients who died during the study,
* Patients who wanted to leave the study,
* Patients who started receiving sedation during the application,
* Patients who added antihypertensive, beta-blocker and similar drugs to their routine treatment during the application,
* Patients who received inotropic treatment (dopamine, steradin and others) during the application,
* Patients who started receiving analgesia treatment during the application,
* Patients who developed ulcers, necrotic tissue and infection at the points where pressure will be applied during the application,
* Patients who started receiving respiratory support from the device during the application,
* Patients who had a Glasgow Coma Scale score of ≤13, mean arterial pressure of ≤65 and SpO2 of ≤85 during the application will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Visual Assessment Scale | 1st day and second day- morning and evening; 15 minutes before application and 30 minutes after the application
  VAS is a measurement tool frequently used in the clinic for pain assessment. The ruler, which is indicated as 0-10 cm or 0-100 mm, has no pain (0) written on one end and the most severe pain (10) on the other end. It is scored between 0-10. The patient marks the point on the ruler where he feels the pain.
Spielberg State-Trait Anxiety Scale | 1st day and second day- morning and evening; 15 minutes before application and 30 minutes after the application and third day morning.
  The scale consists of two sub-dimensions measuring continuous and state anxiety. There are 20 questions for each sub-dimension on a 4-point Likert scale (not at all = 1, a little = 2, a lot = 3, completely = 4). The minimum-maximum score range that can be obtained from the scale varies between 20-80. Increasing scores on the scale indicate an increase in the level of anxiety.
Physiological Parameters Assessment Form | 1st day and second day- morning and evening; 15 minutes before application and 30 minutes after the application
  Systolic Blood Pressure (mm/Hg), Diastolic Blood Pressure (mm/Hg), Respiratory Rate, Heart Rate (Pulse) (beats/min) and Saturation parameters measured before and after acupressure of the intervention and placebo groups will be recorded. Systolic blood pressure measurements will be averaged. Diastolic blood pressure measurements will be averaged. Saturation measurements will be averaged. Respiratory rate measurements will be averaged. Heart Rate (Pulse) measurements will be averaged.
Nursing Presence Scale | 1st day 15 minutes before application and third day morning.
  The scale designed as a 5-point Likert is scored as follows; (never: 1 point), (rarely: 2 points), (occasionally/sometimes: 3 points), (frequently: 4 points) and (always: 5 points). The minimum and maximum scores that can be obtained from the scale are calculated between 24-120. An increase in the score obtained from the scale means that the behaviors in which the patient presents the presence of the nurse have increased and that the patient perceives these behaviors positively.

SECONDARY OUTCOMES:
Richards-Campbell Sleep Scale | 1st day and second day- morning and evening; 15 minutes before application and 30 minutes after the application and third day morning.
  The scale consists of 6 items in total. Each item on the scale is graded between 0 and 100 points. The result is found by dividing the total score obtained from the scale by the number of questions. A score between "0-25" indicates very poor sleep, and a score between "76-100" indicates very good sleep. The minimum score on the scale is calculated as 0, and the maximum score is calculated as 100. An increase in the score obtained from the scale indicates an increase in sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Ozlem Canbolat, Ankara, Turkey (Türkiye)